CLINICAL TRIAL: NCT02173873
Title: Ziv-aflibercept in Eyes With Eyes With Retinal Diseases and Poor Vision-phase I
Brief Title: Ziv-aflibercept in Eyes With Retinal Diseases and Poor Vision-phase I
Acronym: ZIV
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rafic Hariri University Hospital (Other)
Responsible Party: Principal Investigator, Ahmad Mansour, MD, Clinical Professor, AUB, Chair, Department of Opthalmology, Rafic Hariri Hospital, Rafic Hariri University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INV 2014-194
Record Dates: First submitted 2014-06-14; First posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Age Related Macular Degeneration; Central Retinal Vein Occlusion
Keywords: Age related macular degeneration; central retinal vein occlusion
MeSH Terms: conditions — Macular Degeneration; Retinal Vein Occlusion | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- one injection of ziv aflibercept intravitreal route (Experimental): Intervention: Inject 0.05 ml of zaltrap into the vitreous of blind eyes with various diseases (AMD, CRVO) and monitor vision and OCT 1 day and 1 week after injection
  Interventions: Drug: ziv-aflibercept drug

INTERVENTIONS:
Drug: ziv-aflibercept drug — intravitreal injection of ziv-ablicerpt in one eye of each patient with retinal disease and poor vision
  Other Names: Zaltrap

SUMMARY:
Aflibercept is FDA approved and the same molecule is available as hyperosmolar for oncology (cost 800 USD for 4ml) and isoosmolar for Ophthalmology (cost 1,770 USD for 0.05ml injection). The 4ml bottle can be fractionated to be used in 40 patients hence the 0.05 ml injection would cost 20 USD for patients. Animal studies showed the injection is safe, knowing that the rabbit vitreous volume is 3-4 times smaller than the human eye. Our pilot study is to ascertain if the approved molecule for oncology when injected in the eye is safe as it is diluted into 5ml vitreous (100 times dilution). If this is so then we can save the patient 100 times for the most efficient antiVEGF that is used for maculopathy in various diseases (AMD, DME, CRVO, etc..)

DETAILED DESCRIPTION:
Protocol Inject 0.05 ml of zaltrap coumpounded in a sterile way into the vitreous of blind eyes (vision less than 20/100) with various diseases of the retina that require antiVEGF therapy after patient consent. Vision will be monitored 15 minutes, 1 day and 1 week after injection. SD-OCT will be performed before and after 1 week to look for possible side effects.

The safety and efficacy of Eylea in the treatment of macular edema following CRVO3,4 were assessed in 2 randomized, multicenter, double-masked, sham-controlled studies: COPERNICUS and GALILEO. A total of 358 patients were treated and evaluable for efficacy (217 with Eylea) in the two studies. In both, patients were randomly assigned in a 3:2 ratio to either 2 mg Eylea administered every 4 weeks, or sham injections (control group) administered every 4 weeks for a total of 6 injections. After 6 monthly injections, patients continued to receive Eylea treatment during weeks 24 to 52 only if they met pre-specified retreatment criteria (PRN), except for patients in the sham control group in the GALILEO study who continued to receive sham injections through week 52. In the COPERNICUS study, after 6 months, 56% of patients receiving Eylea 2 mg monthly gained at least 15 letters of BCVA from baseline, as measured by ETDRS, compared to 12% of patients receiving sham injections (p<0.01), the primary endpoint of the study. Patients receiving Eylea 2 mg monthly gained, on average, 17.3 letters of vision compared to a mean loss of 4.0 letters with sham control injections (p<0.01), a secondary endpoint.

Ziv-aflibercept or zaltrap6 (Sanofi-Aventis US, LLC, Bridgewater, NJ/Regeneron Pharmaceuticals, Inc, Tarrytown, NY) is FDA approved for the treatment of metastatic colorectal cancer. During Bascom Palmer Eye Institute's Angiogenesis, Exudation, and Degeneration February 2014 conference, Michel Eid Farah, João R. Dias, Fernando M. Penha, and Eduardo B. Rodrigues investigated the safety of ziv-aflibercept in vitro and in vivo. In vitro toxicity was verified using ARPE-19 cultured cells exposed to anti-angiogenic vs balanced salt solution (BSS) for 10 minutes. Viability was assessed by 3-(4,5-dimethylthiazol-2-yl)-2,5-diphenyltetrazolium bromide (MTT) assay, which evaluates cell viability by mitochondrial activity. No signs of cell toxicity were observed, and cell viability was similar for ziv-aflibercept, aflibercept, and BSS. For the in vivo study, they tested 1 injection of 0.05 mL ziv-aflibercept vs aflibercept in the right eyes of 18 rabbits, 9 eyes in each group. BSS was injected in the fellow eyes and served as control. After the injections, all animals were examined by funduscopy, SD-OCT), and ERG at baseline, 24 hours, and 7 days. Aqueous, vitreous, and serum samples were collected at baseline, 24 hours, and 7 days for pH and osmolarity analysis. The animals were sacrificed and the eyes were enucleated for morphologic study by light and electron microscopy. No abnormalities were found at 24 hours or 7 days after intravitreal injection of either drug when assessed by fundus exam and SD-OCT, ERG, and histology as well as transmission microscopy. There were also no changes in osmolarity in the aqueous humor or vitreous samples in any group after 24 hours and 1 week.

ELIGIBILITY:
Inclusion Criteria: Eyes with wet age related macular degeneration, central retinal vein occlusion or diseases that require antiVEGF especially in poor vision eyes -

Exclusion Criteria: eyes that had recent eye surgery, inability to sign consent, blepharitis, conjunctivitis

-

Ages: 16 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Ziv-aflibercept in retinal diseases with poor vision: Safety monitoring by OCT and visual acuity | 2 years
  anterior chamber, vitreous, lens, retina exam PLUS OCT and visual acuity
OCT retinal structure | 2 years
  OCT, visual acuity measure, inflammation measure

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Mansour, MD, Study Chair — RHUH
Locations (1):
- Rafic Hariri University Hospital, Beirut, Lebanon

REFERENCES:
- [Background] Malik D, Tarek M, Caceres del Carpio J, Ramirez C, Boyer D, Kenney MC, Kuppermann BD. Safety profiles of anti-VEGF drugs: bevacizumab, ranibizumab, aflibercept and ziv-aflibercept on human retinal pigment epithelium cells in culture. Br J Ophthalmol. 2014 Jun;98 Suppl 1(Suppl 1):i11-16. doi: 10.1136/bjophthalmol-2014-305302. PMID 24836865
- [Derived] Mansour AM, Al-Ghadban SI, Yunis MH, El-Sabban ME. Ziv-aflibercept in macular disease. Br J Ophthalmol. 2015 Aug;99(8):1055-9. doi: 10.1136/bjophthalmol-2014-306319. Epub 2015 Feb 12. PMID 25677668
- See also: Safety profiles of anti-VEGF drugs: bevacizumab ... www.ncbi.nlm.nih.gov/pubmed/24836865 — http://www.ncbi.nlm.nih.gov/pubmed/24836865